CLINICAL TRIAL: NCT06512597
Title: Combination Therapy of Resilience Intervention With Biologics in Crohn's Disease (CATHARSIS Trial)
Brief Title: Behavioral Therapy for Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Laurie Keefer, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-24-00338
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Time

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary Intervention for Combination Therapy - IBD Coping Strategies Program (Experimental): This 7-session protocol is based on Dr. Keefer's validated Project Management for Crohn's disease treatment manual. The program specifically focuses on reducing stress, building resilience, fostering self-confidence and disease acceptance, all of which have been associated with improved adjustment to disease and better self-management outcomes in CD.
  Interventions: Behavioral: Primary Intervention for Combination Therapy - IBD Coping Strategies Program
- Time and Attention Control Group - IBD Support Program (Standard Therapy) (Sham Comparator): This 7-session condition will serve as a Time and Attention Control to the Coping Strategies Program. The therapist will follow Dr. Keefer's previously validated control condition manual focused on supportive listening, disease education and self-reflection.
  Interventions: Behavioral: Time and Attention Control - IBD Support Program

INTERVENTIONS:
Behavioral: Primary Intervention for Combination Therapy - IBD Coping Strategies Program — psychosocially credible treatments each comprised of seven 45-minute sessions over a 12-week period, delivered via telemedicine.
  Arms: Primary Intervention for Combination Therapy - IBD Coping Strategies Program
Behavioral: Time and Attention Control - IBD Support Program — psychosocially credible treatments each comprised of seven 45-minute sessions over a 12-week period, delivered via telemedicine.
  Arms: Time and Attention Control Group - IBD Support Program (Standard Therapy)

SUMMARY:
People living with Crohn's disease (CD) experience psychological and emotional symptoms, in addition to known chronic and disabling physical symptoms, which prevent them from living their life to the fullest (flourishing). Depression and anxiety are experienced by 30% of people living with CD and 60% of inflammatory bowel disease (IBD) patients continue to report chronic pain, stress, sleeplessness, and fatigue, even when they are "objectively" in remission. Psychological stress has been endorsed by 70% of patients with IBD as a key trigger for disease activity which is not surprising given the significance of the gut-brain-microbiome axis, the close communication between the enteric and autonomic nervous systems, and the role of the hypothalamic-pituitary axis and its neuroendocrine and immune functions in the expression of GI symptoms. Interestingly, up to 85% of patients with CD also endorse the positive impact of effective coping skills on disease course. The PI's prior work has suggested that early provision of effective coping strategies, offered at the time of diagnosis or more precisely, immediately prior to biologic medication initiation, could potentially result in faster healing and improved well-being, likely through the combination of 1) physiological mitigation of the stress response and optimization of the gut-brain-microbiome axis; and 2) promotion of effective coping and disease self-management behaviors that promote psychological flourishing despite disease. Unfortunately, to date, early effective psychosocial care has been limited by concerns over reimbursement for psychological services, access to qualified IBD mental health professionals, and the lack of a standardized methodology focused on the brain-gut stress response and how to assess, monitor, communicate and maintain tight control over both physical and emotional well-being. CATHARSIS is a rigorous, placebo-controlled, randomized controlled trial of coping strategies plus medication for 170 people living with Crohn's for less than 5 years who are about to start a new biologic medication due to active disease. Outcomes include improvements in emotional well-being as well as clinical and endoscopic remission over a 12-month period. The overall goal of the study is to demonstrate that it is essential to combine biologic therapy and psychosocial care to ensure optimal and long-term positive outcomes in CD.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years old) of any sex, gender, and racial/ethnic background with an endoscopically and histologically confirmed CD diagnosis will be eligible.
* Participants must have active CD symptoms as defined by a Crohn's Disease Activity Index (CDAI) of at least 220 and
* Active endoscopic inflammation defined as a Simple Endoscopic Score for CD (SES-CD) > 6 (or ≥4 for isolated ileal disease) on most recent colonoscopy OR active disease on imaging study OR elevated calprotectin/CRP levels
* Must be planning to start an anti-TNF (adalimumab, certolizumab, or infliximab) or anti-IL-23 (risankizumab, guselkumab, mirikizumab) within the prior 2 weeks or in the next 6 weeks.
* Participants will need to live in one of Dr Keefer's 30+ PSYPACT licensed states.

Exclusion Criteria:

* Endoscopically inactive Crohn's disease at baseline.
* Unable to consent to participation.
* Pregnant or planning to become pregnant in next 12 months.
* Severe psychiatric symptoms.
* Surgical history for CD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
The PROMIS Global Health Scale | at week 24
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale
  A series of person-centered measures that evaluate and monitor physical, mental, and social health in adults and children. 10-item patient-reported questionnaire. standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.

SECONDARY OUTCOMES:
Psychological Well-Being Scale | at weeks 12, 24, 36 and 52
  Each item uses a 7-point scale (1=strongly agree; 7=strongly disagree) There are 6 subscales: The Autonomy subscale, The Environmental Mastery subscale, The Personal Growth subscale, The Positive Relations with Others subscale, The Purpose in Life subscale, and The Self-Acceptance subscale.
  Subscales scored from 3 to 21, with higher score indicating higher levels of psychological well-being.
  Full scale from 18 to 126, with higher score indicating higher levels of psychological well-being.
Inflammatory Bowel Disease Self-Efficacy Scale (IBD-SES) | at weeks 12, 24, 36 and 52
  The IBD-SES is a 13-item questionnaire. Each item scored 1 (completely disagree) to 5 (completely agree). The IBD-SES assesses how patients manage things related to their IBD and other things in their everyday life. For each statement, they must select the number that best fits the answer for the past two weeks. Full scale from 13-65 with higher score indicating better health outcomes.
NIH PROMIS-29 | at weeks 12, 24, 36 and 52
  Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) measures seven domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and the ability to participate in social roles and activities. Each domain has 4 questions ranked on a 5-point scale, and refer to the 7 previous days except physical function which has not time frame.
  Scoring is standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points.
  Higher scores indicate poorer health outcomes for anxiety, depression, fatigue, ability to participate in social roles and activities, and pain interference domains.
  Lower scores reflect worse outcomes for physical function and sleep disturbances domains.
Crohn's Disease Activity Index (CDAI) | at weeks 12, 36, and 52
  Crohn's Disease Activity Index (CDAI) score is a measurement of the severity of the Crohn's disease symptoms. Full scale ranges from 0-600, with higher score indicating more severe disease.
Patient-Reported Outcomes (PRO2) | at weeks 12, 24, 36, and 52
  The PRO2 questionnaire assesses stool frequency and rectal bleeding, each question scored from 0-3. Full scale from 0-6, with higher score indicating poorer health outcomes.
Inflammatory Bowel Disease Questionnaire (IBDQ) | at weeks 12, 24, 36, and 52
  Inflammatory Bowel Disease Questionnaire (IBDQ) is a 32 item questionnaire. Full scale from 32-224, with higher score indicating better quality of life.
UCLA GI Symptom Severity Score | at weeks 12, 24, 36, and 52
  UCLA GI Symptom Severity Score rates overall severity of GI symptoms. Full scale from 0-20, with higher score indicating more intense symptoms.
Simple Endoscopic Score for Crohn's Disease (SES-CD) | at 24 weeks
  Simple Endoscopic Score for Crohn's Disease (SES-CD) is used to quantify and compare inflammatory load. The Simple Endoscopic Score for Crohn Disease (SES-CD) assesses the size of mucosal ulcers, the ulcerated surface, the endoscopic extension and the presence of stenosis. Each item is scored from 0-3, with total score from 0-60. Higher score indicates poorer health.
C-reactive protein level | up to 24 weeks
  C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation in the body. It is one of a group of proteins, called acute phase reactants that go up in response to inflammation. The levels of acute phase reactants increase in response to certain inflammatory proteins called cytokines. These proteins are produced by white blood cells during inflammation.
  The CRP test is a general test to check for inflammation in the body. It is not a specific test. This means it can reveal inflammation somewhere in the body, but it cannot pinpoint the exact location or reason.
fecal calprotectin level | up to 24 weeks
  Inflammatory markers measured in stool samples can be used for assessing the disease in patients who have undergone surgery. A stool test called fecal calprotectin can be of help in determining if symptoms are indicative of a flare-up of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Keefer, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Ryan Ungaro, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Gastroenterology Associates, New York, New York

IPD SHARING:
Plan to Share IPD: No